CLINICAL TRIAL: NCT02420574
Title: Assessment of Drug Efficacy of Albendazole Bought on Local Market Against Soil-transmitted Helminth Infections in School Children in Jimma, Ethiopia
Brief Title: Assessment of Drug Efficacy of Local Albendazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B670201319330
Record Dates: First submitted 2015-03-26; First posted 2015-04-20 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Helminthiasis
MeSH Terms: conditions — Helminthiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALB-BENDEX (Active Comparator): albendazole, 400 mg, single oral dose, (BENDEX)
  Interventions: Drug: albendazole BENDEX
- ALB-OVIS (Active Comparator): albendazole, 400 mg, single-oral dose, (OVIS)
  Interventions: Drug: albendazole OVIS

INTERVENTIONS:
Drug: albendazole BENDEX — randomized clinical trial with 2 parallel arms
  Other Names: BENDEX/OVIS
  Arms: ALB-BENDEX
Drug: albendazole OVIS
  Arms: ALB-OVIS

SUMMARY:
Infections with soil-transmitted helminthes (STH) occur throughout the developing world and remain a major public health problem in the poorest communities. Preventive chemotherapy (PC) programs in which single-dose albendazole 400 mg or single-dose mebendazole 500 mg - the drugs of choice for STH - are administered at the population level, is the main strategy for STH control. To ensure quality, these drugs are being widely donated by GlaxoSmithKline (GSK) (albendazole (ALB), Zentel) and Johnson & Johnson (mebendazole (MEB), Vermox). In addition to this, there are a wide variety of ALB and MEB tablets available on the local market. Although little is known about the quality of anthelmintics sold for human use, several publications have reported variability in the quality of generic anthelmintics used in veterinary medicine. The main objective of the present study is to compare the efficacy of two ALB brands bought on the local market, including OVIS (Korea, DAEHWA pharmaceutical) and BENDEX (India, Cipla)

DETAILED DESCRIPTION:
1. Background Infections with soil-transmitted helminthes (STH) occur throughout the developing world and remain a major public health problem in the poorest communities. Infection is caused by four main species of worms commonly known as roundworms (Ascaris lumbricoides), whipworms (Trichuris trichiura) and hookworms (Ancylostoma duodenale and Necator americanus). It is estimated that STH affects more than 2 billion people worldwide, of which 450 million have significant morbidity attributable to their infection, and hence are one of the most important neglected tropical diseases. Children and pregnant women are the two most vulnerable groups. Children experience growth stunting and diminished physical fitness as well as impaired memory and cognition, resulting in impaired childhood educational performance and reduce school attendance; pregnant women suffer significant morbidity with hookworm-associated anemia likely contributing to maternal mortality.

   Preventive chemotherapy (PC) programs in which single-dose albendazole 400 mg or single-dose mebendazole 500 mg - the drugs of choice for STH - are administered at the population level, is the main strategy for STH control. To ensure quality, these drugs are being widely donated by GlaxoSmithKline (GSK) (albendazole (ALB), Zentel) and Johnson & Johnson (mebendazole (MEB), Vermox). In addition to this, there are a wide variety of ALB and MEB tablets available on the local market. Although little is known about the quality of anthelmintics sold for human use, several publications have reported variability in the quality of generic anthelmintics used in veterinary medicine. The concentrations of nine anthelmintic products (levamisol and MEB) purchased in pharmacies and from agricultural merchants in Kenya varied from 0 to 118 % of their claimed composition. Efficacy studies of seven brands of ALB against gastrointestinal nematodes in sheep in Ethiopia showed that the efficacy of only five of the seven brands was satisfactory.
2. Objectives The main objective of the present study is to compare the efficacy of two ALB brands bought on the local market, including OVIS (Korea, DAEHWA pharmaceutical) and BENDEX (India, Cipla)
3. Materials and methods 3.1. Study Population School children between 4 and 18 years old are the focus of this study because of two main reasons: school children are normally a major target for regular treatment with anthelminthic, because they are the group that usually has the heaviest worm burdens for A. lumbricoides and T. trichiura, and are steadily acquiring hookworm infections. In addition, they are in a period of intense physical and intellectual growth. Deworming schoolchildren has a considerable benefit on their nutritional status, physical fitness, appetite, growth and intellectual development.

   3.2. Study design The study design is based on the recent WHO guidelines on how to assess drug efficacy against STH. Briefly, following obtaining informed consent, school children in the target age range group will be recruited and asked to provide a recent stool sample (an interval of less than 4 hours) that will be processed to determine the fecal egg counts (FEC) for each STH present. For the initial sampling the aim is to enroll at least 650 children. This is based on a sample size of at least 50 infected subjects for each STH in each treatment arm (cfr WHO guidelines), an apparent prevalence of 20% for the least prevalent STH species and a drop out of 20%.

   All children providing stool samples will be randomized across two treatment arms. Fourteen days after treatment a second fecal sample will be collected from the children to determine again FEC. Subjects who are unable to provide a stool sample at follow-up, or who are experiencing a severe concurrent medical condition or have diarrhea at time of the first sampling, will be excluded from the study. At follow-up all students will receive a single oral dose ALB tablet that was donated by GSK through WHO (Zentel).

   3.3. Determination of FEC of STH All fecal samples will be processed using the McMaster egg counting technique (analytic sensitivity of 50 EPG) for the detection and the enumeration of infections with A. lumbricoides, T. trichiura and hookworms.

   3.4. Statistical analysis The efficacy of the brands against each of the three STH will be measured by reduction in FEC using the formula below.

   The efficacy of the drugs will be classified into 'satisfactory', 'doubtful' and 'reduced' using the criteria summarized in Table 1.

   Table 1. The criteria based on FECR classifying efficacy of drugs into 'satisfactory', 'doubtful' and 'reduced' A. lumbricoides T. trichiura Hookworm Satisfactory FECR ≥ 95% FECR ≥ 50% FECR ≥ 90% Doubtful 95%> FECR ≥95% 50%> FECR ≥40% 90%> FECR ≥80% Reduced FECR ≤85% FECR ≤40% FECR ≤80%

   3.5. Interpretation In any case of doubtful or reduced efficacy further steps will be taken to assess the efficacy of the drug.
4. Ethical issues This study will be reviewed by the Ethics committees of the Faculty of Medicine, Ghent University (Belgium) and the Jimma University, Jimma (Ethiopia).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 5-18 years old.
2. Sex: males and females.
3. Signed of written informed consent sheet by parents/or guardians, and those who volunteered to comply with study procedures (stool submission, drug treatment).
4. Females: was not pregnant (as verbally assessed by clinician upon enrolled to treatment).

Exclusion Criteria:

1. Had vomit within 4 hours after drug administration.
2. Had diarrhea at time of the first sampling.
3. Subjects who were unable to provide a stool sample at follow-up,
4. Subjects who experienced a severe concurrent medical condition
5. Subjects with known history of allergic reaction to ALB.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 679 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Egg reduction rate | 14 days after administration of the drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Vercruysse, PhD, Principal Investigator — University Ghent

REFERENCES:
- [Background] Bethony J, Brooker S, Albonico M, Geiger SM, Loukas A, Diemert D, Hotez PJ. Soil-transmitted helminth infections: ascariasis, trichuriasis, and hookworm. Lancet. 2006 May 6;367(9521):1521-32. doi: 10.1016/S0140-6736(06)68653-4. PMID 16679166
- [Background] Bundy DA, Hall A, Medley GF, Savioli L. Evaluating measures to control intestinal parasitic infections. World Health Stat Q. 1992;45(2-3):168-79. PMID 1462652
- [Background] Crompton DW, Nesheim MC. Nutritional impact of intestinal helminthiasis during the human life cycle. Annu Rev Nutr. 2002;22:35-59. doi: 10.1146/annurev.nutr.22.120501.134539. Epub 2002 Jan 4. PMID 12055337
- [Background] Curtale F, Pokhrel RP, Tilden RL, Higashi G. Intestinal helminths and xerophthalmia in Nepal. A case-control study. J Trop Pediatr. 1995 Dec;41(6):334-7. doi: 10.1093/tropej/41.6.334. PMID 8606439
- [Background] De Clercq D, Sacko M, Behnke J, Gilbert F, Dorny P, Vercruysse J. Failure of mebendazole in treatment of human hookworm infections in the southern region of Mali. Am J Trop Med Hyg. 1997 Jul;57(1):25-30. doi: 10.4269/ajtmh.1997.57.25. PMID 9242313
- [Background] Monteiro AM, Wanyangu SW, Kariuki DP, Bain R, Jackson F, McKellar QA. Pharmaceutical quality of anthelmintics sold in Kenya. Vet Rec. 1998 Apr 11;142(15):396-8. doi: 10.1136/vr.142.15.396. PMID 9586132
- [Background] Nokes C, Bundy DA. Does helminth infection affect mental processing and educational achievement? Parasitol Today. 1994 Jan;10(1):14-8. doi: 10.1016/0169-4758(94)90348-4. PMID 15275558
- [Background] Stephenson LS, Latham MC, Adams EJ, Kinoti SN, Pertet A. Physical fitness, growth and appetite of Kenyan school boys with hookworm, Trichuris trichiura and Ascaris lumbricoides infections are improved four months after a single dose of albendazole. J Nutr. 1993 Jun;123(6):1036-46. doi: 10.1093/jn/123.6.1036. PMID 8505663
- [Background] Stoltzfus RJ, Albonico M, Chwaya HM, Savioli L, Tielsch J, Schulze K, Yip R. Hemoquant determination of hookworm-related blood loss and its role in iron deficiency in African children. Am J Trop Med Hyg. 1996 Oct;55(4):399-404. doi: 10.4269/ajtmh.1996.55.399. PMID 8916795
- [Background] Vercruysse J, Behnke JM, Albonico M, Ame SM, Angebault C, Bethony JM, Engels D, Guillard B, Nguyen TV, Kang G, Kattula D, Kotze AC, McCarthy JS, Mekonnen Z, Montresor A, Periago MV, Sumo L, Tchuente LA, Dang TC, Zeynudin A, Levecke B. Assessment of the anthelmintic efficacy of albendazole in school children in seven countries where soil-transmitted helminths are endemic. PLoS Negl Trop Dis. 2011 Mar 29;5(3):e948. doi: 10.1371/journal.pntd.0000948. PMID 21468309
- See also: World Health Organization (2005) Deworming for health and development. Report of the third global meeting of the partners for parasitic control. WHO/CDS/CPE/PVC/2005.14, World Health Organization, Geneva. — http://whqlibdoc.who.int/hq/2005/who_cds_cpe_pvc_2005.14.pdf
- See also: 6. Kumsa, B., Debela, E., Megersa, B., 2010. Comparative efficacy of albendazole, tetramisole and ivermectin against gastrointestinal nematodes in naturally infected goats in Ziway, Oromia Regional State (Southern Ethiopia). J Anim Vet Adv 9, 2905-2911. — http://medwelljournals.com/abstract/?doi=javaa.2010.2905.2911